CLINICAL TRIAL: NCT04340635
Title: Analysis of Eye Bioparametric Data of Chinese Population Based on Big Data
Brief Title: Multi-center Ocular Biological Parameters Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHIRB2018020
Record Dates: First submitted 2020-03-29; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Cataract
Keywords: Corneal astigmatism; axial length (AL), anterior chamber depth (ACD); partial coherence interferometry
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multi-center data collection: Without intervention

INTERVENTIONS:
Other:  — Without intervention

SUMMARY:
This study is a multi-center study, which collects data from multiple regions to obtain the general biological characteristics of the Chinese population. The formula for calculating the artificial lens power based on foreign populations is effectively modified based on the Chinese population.

DETAILED DESCRIPTION:
①Relevant domestic studies on the biological characteristics of the eye are mainly limited to a certain city and region. Most of the studies that represent the biological characteristics of the general population in China and the differences in biological parameters at home and abroad are in the research process, or Semi-finished products.

②The investigators found in clinical observation that the eyeball biological data of the Chinese population may not be consistent with the foreign population.

③ This study is the first study of human eye biological parameters based on different regions of large-scale populations in China, which is of great significance for understanding the human eye structure in different regions of China.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 50 years

Exclusion Criteria:

* history of refractive surgery,
* corneal diseases
* ocular inflammation
* trauma

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Select elderly cataract patients from different regions of China (at least one representative city in each of east, south, west, north, and central China) who were treated in Aier Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
axial length (AL) | 1 hour
  Measured using the partial coherence laser interferometry (IOLMaster, Carl Zeiss Meditec, Germany)
anterior chamber depth (ACD) | 1 hour
  Measured using the partial coherence laser interferometry (IOLMaster, Carl Zeiss Meditec, Germany)
keratometric power (K) | 1 hour
  Measured using the partial coherence laser interferometry (IOLMaster, Carl Zeiss Meditec, Germany)
corneal astigmatism (CA) | 1 hour
  Measured using the partial coherence laser interferometry (IOLMaster, Carl Zeiss Meditec, Germany)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Aier Eye Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qian Z, Xie X, Yang J, Ye H, Wang Z, Chen J, Liu H, Liang J, Jiang L, Zheng C, Chen X. Detection of shallow anterior chamber depth from two-dimensional anterior segment photographs using deep learning. BMC Ophthalmol. 2021 Sep 22;21(1):341. doi: 10.1186/s12886-021-02104-0. PMID 34551738